CLINICAL TRIAL: NCT04864483
Title: Sahoor Meal Regimen for Patients With Type1 Diabetes; Randomized Cross Over Design of Two Regimens
Brief Title: Sahoor Meal Regimen for Patients With Type1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah International Medical Research Center (Other)
Responsible Party: Principal Investigator, Reem Mohammad Alamoudi, CONSULTANT ENDOCRINOLOGY, King Abdullah International Medical Research Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RJ20/446/J,
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Type1diabetes; Fasting Hypoglycemia
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Intervention Model Description: Randomized cross over design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early sahoor with predawn snack (Experimental): To take the Sahoor meal 1:30-2 hours before dawn with insulin dose then a pre-dawn snack with no insulin
  (Sahoor is the latest meal before starting the fast at dawn during the month of Ramadan. The intervention is meal timing in relation to start of fast and does not involve any medications).
  Interventions: Other: Meal timing in relation to time of starting the fast
- Late Sahoor meal (within 30 minjted of dawn) with insulin dose (Experimental): To take sahoor meal as late as possi le with usual insulin dose
  (Sahoor is the latest meal before starting the fast at dawn during the month of Ramadan. The intervention is meal timing in relation to start of fast and does not involve any medications).
  Interventions: Other: Meal timing in relation to time of starting the fast

INTERVENTIONS:
Other: Meal timing in relation to time of starting the fast — as described

SUMMARY:
To examine effects of two approaches to sahoor meal consumption during Ramadan on blood sugar control and incidence of early day hypoglycemic episodes requring the discontinuation of fasting.

DETAILED DESCRIPTION:
Most studies and guidelines regarding insulin dose adjustments have focused on basal insulin modification rather than boluses or timing of meals. There hasn't been so far any study that examines a specific dose reduction or timing that is best to avoid early day (post Suhoor) hypo or hyperglycemia, and the advised dose reductions are based on expert opinion with small observational studies that used certain dose changes.

The timing of sleep and meals are different during Ramadan and therefore have a direct impact on blood glucose levels, we demonstrated in a previous prospective cohort of 156 T1DM patients contrary to other studies, the post suhoor and early day period had the highest incidence time for hypoglycemia in the Saudi population. It is therefore necessary to understand how adjustments to the timing of the meals and their doses can achieve better glycemic control during fastin Ramadan. Current guidelines recomend that the Suhoor meal is delayed as much as possible in order to reduce the fasting duration to be taken with a claculated insulin dose. However, the concern is that this would not allow patients to correct the hypoglycemic or hyperglycemic events related to miscalculation of Suhoor insulin dose if they occur as the fasting time begins and they must break their fast to correct their blood glucose levels. Many people with T1DM do not count meal carbohydrates correctly, therefore, there is a need for an approach that allows patients to correct their blood glucose levels after having a large meal that requires insulin administration without having to break their fast, as well as the ability to have a snack or a late Suhoor without the need for insulin administration to minimize the fasting period and insure that the blood glucose is in range before starting to fast. The approach that we are proposing will allow patients to do that by having the Suhoor meal with its bolus at least two hours before fasting begins, and having a low carbohydrate snack - late suhoor- just before starting to fast without the need for insulin administration (regimen 1). It is going to be compared with having the Suhoor with its insulin bolus just before the start of fasting (regimen 2).

ELIGIBILITY:
Inclusion Criteria:

1. DM type 1
2. Age > 14 years
3. Diagnosis of type 1 DM of more than 6 months.
4. Committed to do SMBG or on CGM
5. On Multiple Daily Injections or insulin pumps
6. On carbohydrate counting for meal dosing
7. Have previously fasted Ramadan
8. Are willing to fast this year
9. Well educated about requirements for fasting Ramadan

Exclusion Criteria:

1. Cognitive impairment or learning disability
2. Renal and hepatic impairment
3. Adrenal insufficiency
4. Pregnancy
5. Alcohol consumption
6. Any diagnosed psychiatric disease

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-03-21 (Actual); Primary Completion 2021-06-27 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Incidence of early day hypoglycemia | 1 month
  To determine if taking insulin dose suhoor meal 90 minutes before dawn plus a predawn high protein snack is associated with less rates of hypoglycemia -(we will consider glucose level of 70 mg/dl ( 3.9 mmol/l) and below as the level of hypoglycemia - compared to taking insulin dose suhoor meal 15-30 minutes before dawn during fasting Ramadan in patietnts with T1DM on MDI or insulin pump

SECONDARY OUTCOMES:
number of days fasting discontinued | 1 month
  To estimate the difference between the two regimens in number of days they needed to brake their fast
Hyperglycemia incidence during fasting | 1 month
  To estimate the difference between the two regimen in daytime hyperglycemia
Blood sugar control | 1 month
  To assess the difference in glycemic control between the two regimens using estimated A1c
Incidence of complications | 1 month
  To estimate the difference between the two groups in rate of severe hyperglycemia and /or DKA
Glucose variability | 1 month
  To estimate the difference between the two regimens in glucose variability
Patient satisfaction and preference | 1 month
  To estimate the difference between the two regimens in patients' preferences

CONTACTS AND LOCATIONS:
Overall Officials: Reem M Alamoudi, Principal Investigator — King Abdullah International Medical Research Center
Locations (1):
- KingAbullahIMRC, Jeddah, Western, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided